CLINICAL TRIAL: NCT04330001
Title: Exploratory Clinical Study for Techniques Associated With the Fluid Accommodating IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ILR286-E003
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Aphakia; Presbyopia
Keywords: IOL; Cataract; Accommodation
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- FAIOL (Experimental): Implantation of FAIOL in the capsular bag in the posterior chamber of the eye. The IOL is intended to be used over the lifetime of the subject.
  Interventions: Device: Alcon Fluid Accommodating Intraocular Lens; Other: Top Con Autorefractor

INTERVENTIONS:
Device: Alcon Fluid Accommodating Intraocular Lens — Intraocular lens intended to treat presbyopia by dynamically adjusting power, resulting in a continuous range of vision from distance to near.
  Other Names: FAIOL; FluidVision MX Accommodating IOL
Other: Top Con Autorefractor — Device intended to automatically determine the focusing characteristics of the eye

SUMMARY:
The purpose of this clinical study is to assess the repeatability of objective refraction using auto refraction on subjects bilaterally implanted (implanted in both eyes) with the Fluid Accommodating IOL (FAIOL).

DETAILED DESCRIPTION:
Subjects will be expected to attend 10 office visits from screening to exit. The total expected duration of participation for each subject in this study is approximately 12 months. The second eye surgery will take place within 7-15 days from the date of the first implanted eye. The primary endpoint will be collected at Month 1, following the 2nd eye implant date.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend all scheduled study visits as required per protocol
* 22 years of age or older
* Bilateral cataracts
* Corneal astigmatism ≤ 1.25 D
* Clear intraocular media other than cataract
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential, defined as all women who are physiologically capable of becoming pregnant and who are not postmenopausal for at least 1 year or are less than 6 weeks since sterilization, are excluded from participation if any of the following apply:

  1. are currently pregnant,
  2. have a positive urine pregnancy test result at V0,
  3. intend to become pregnant during the study period,
  4. are breast-feeding.
* Subjects taking medications that may affect accommodation, confound the outcome, or as per the Investigator's opinion may increase the risk to the subject
* Glaucoma
* Significant corneal or retinal abnormalities, per the Investigator's opinion, or other disease or pathology other than cataract expected to reduce postoperative vision
* Monocular patient, significant permanent visual function loss, or binocular vision anomalies as evaluated by specific testing
* Previous corneal procedure (such as LASIK, keratotomy, LRI) or plans to have additional corneal procedures during the study
* Systemic disease that could increase the operative risk or confound the outcome
* Other protocol-specified exclusion criteria may apply

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Repeatability of objective refraction | Month 1 (post 2nd eye implant)
  Two assessments of objective refraction (sphere, cylinder, and spherical equivalent) using auto refraction will be made on the same day. Repeatability of objective refraction will be evaluated using the Intra-class correlation coefficient (ICC), separately by eye. ICC is evaluated as the proportion of all variation that is not due to measurement error. Higher values of ICC indicate lower error variance and hence better repeatability. Repeatability of objective refraction will be assessed with and without cycloplegia (temporary paralysis of the ciliary muscle).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operation Lead CDMA Surgical, Study Director — Alcon Research
Locations (2):
- Alcon Investigator 8071, San Salvador, El Salvador
- Alcon Investigator 8165, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No